CLINICAL TRIAL: NCT05169619
Title: Epi-Asthma: Prevalence and Characterisation of Asthma Patients According to Disease Severity in Portugal
Brief Title: Prevalence and Characterisation of Asthma Patients According to Disease Severity in Portugal
Acronym: Epi-Asthma
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Faculdade de Medicina da Universidade do Porto - CINTESIS (Unknown); Universidade do Minho - ICVS (Unknown)
Responsible Party: Sponsor
Other Study IDs: D2287R00155
Record Dates: First submitted 2021-11-15; First posted 2021-12-27 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Asthma
Keywords: Asthma; Severe Asthma; Difficult-to-treat asthma; Prevalence
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine the prevalence of Asthma, Difficult-to-Treat and Severe Asthma in Portugal, and characterize patients to better understand their disease characteristics, treatment profile and health care resource use to improve clinical management of the disease.

DETAILED DESCRIPTION:
Data on the epidemiology of asthma in Portugal were mainly grounded in studies using questionnaires and covering limited age groups. Studies assessing the prevalence of asthma diagnosis and of its sub-groups with more accurate methods are therefore needed This study aims to determine the prevalence of asthma, difficult-to-treat and severe asthma in Portugal, and to characterize patients to better understand their disease characteristics, treatment profile and health care resource use to improve clinical management of the disease.

We will conduct a population-based nationwide study with a multicentre stepwise approach, enrolling 7500 adult subjects, randomly selected, from the Portuguese National Health Service patients' database of 38 primary care centres:

STAGE 0 - Phone call invitation and enrolment of participants STAGE 1 - Telephone interview survey to assess respiratory symptoms. STAGE 2 - Clinical assessment, diagnostic confirmation, and patient characterization STAGE 3 - Characterization of asthma patients (sub-group) and characterization of difficult- to-treat asthma & severe asthma patients after 3 months follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Adults =>18 years old registered in Portuguese National Health service patients' database of primary care units.
* Give voluntary signed informed consent,
* Ability to understand ans answer questionnaires.

Exclusion Criteria:

* Participants that have a physical condition that could interfere with the study assessments or prevent the participant from adequately participating in the study (e.g. mobility problems, not able to perform spirometry,…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of study will be adult (=> 18 years) persons registered in the Portuguese National health service patients' database.
  Participants will be enrolled in the study according to proportionate allocation from primary care health units that will be identified based on demographic stratification (i.e. NUTS III)
Sampling Method: Probability Sample
Enrollment: 842 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with asthma, difficult-to-treat asthma, and severe asthma | From date of inclusion until the end of the study currently planned (2,5 years)
  Ratio between the total number of participants with confirmed asthma, difficult-to-treat asthma, and severe asthma and the total number of participants

SECONDARY OUTCOMES:
Subject's characteristics - Age | From date of inclusion until the end of the study currently planned (2,5 years)
  Years
Subject's characteristics - Living in a city or rural community | From date of inclusion until the end of the study currently planned (2,5 years)
  Postal code
Subject's characteristics - Family history | From date of inclusion until the end of the study currently planned (2,5 years)
  Family history of asthma and asthma death and type of relationship
Subject's characteristics - Comorbidities and allergies | From date of inclusion until the end of the study currently planned (2,5 years)
  List of comorbidities with major impact on asthma outcomes
Subject's characteristics - Obesity | From date of inclusion until the end of the study currently planned (2,5 years)
  WHO classification of body mass index
Subject's characteristics - Physical activity | From date of inclusion until the end of the study currently planned (2,5 years)
  Using the brief physical activity assessment questionnaire. This brief physical activity assessment has only two questions and subjects are scored on < 4 (Insufficiently" active) and ⩾4 ("Sufficiently" active).
Subject's characteristics - Health related quality of life | From date of inclusion until the end of the study currently planned (2,5 years)
  Using mini AQLQ Questionnaire AQLQ is a multiple-choice questionnaire for patients with asthma, each choice is assigned a score 1-7. There are 15 questions to answer. The total score is calculated and ranges between 15 and 105. Lower scores indicate worse quality of life.
Subject's characteristics - Healthcare resource use and costs | From date of inclusion until the end of the study currently planned (2,5 years)
  a) Direct resources will include number of inpatient admissions, emergency and hospital visits, medical appointments, diagnostic tests previously performed for asthma treatment in the last 12 months. b) Indirect resources will include reduced productivity of Asthma patients through an ad-hoc questionnaire about absenteeism (work and school days lost because of asthma) and presenteeism (reduced productivity due to asthma) in the last 12 months.
Subject's characteristics - Referral | From date of inclusion until the end of the study currently planned (2,5 years)
  number of patients that should be referral for asthma specialist hospital Consultation or that were referred to Severe Asthma consultation
Disease Characteristics - Age of Asthma onset | From date of inclusion until the end of the study currently planned (2,5 years)
  Age of Asthma onset
Disease Characteristics - Asthma symptoms | From date of inclusion until the end of the study currently planned (2,5 years)
  According to Control of Allergic Rhinitis and Asthma Test (CARAT). CARAT is a 10-item validated Portuguese questionnaire, which allows for the simultaneous assessment of allergic rhinitis and asthma (ARA) control. A score above 24 (min. 0; max. 30) identifies controlled asthma.
Disease Characteristics - Pulmonary function tests | From date of inclusion until the end of the study currently planned (2,5 years)
  Spirometry and reversibility testing
Disease Characteristics - Inflammatory biomarkers | From date of inclusion until the end of the study currently planned (2,5 years)
  Fractional exhaled nitric oxide (FeNO) test and blood eosinophil and neutrophil count,
Disease Characteristics - Exacerbations | From date of inclusion until the end of the study currently planned (2,5 years)
  Number of exacerbations in the past year
Disease Characteristics - Emergency room (ER) visits | From date of inclusion until the end of the study currently planned (2,5 years)
  Number of visits to emergency room (ER) within the past year
Disease Characteristics - Hospital admissions | From date of inclusion until the end of the study currently planned (2,5 years)
  Number of hospital admissions and mean length of hospital stay in the past year
Disease Characteristics - Disease control | From date of inclusion until the end of the study currently planned (2,5 years)
  According to Control of Allergic Rhinitis and Asthma Test (CARAT). CARAT is a 10-item validated Portuguese questionnaire, which allows for the simultaneous assessment of allergic rhinitis and asthma (ARA) control. A score above 24 (min. 0; max. 30) identifies controlled asthma.
Treatment Patterns - Treatment profile (current and last year) | From date of inclusion until the end of the study currently planned (2,5 years)
  Stage of GINA treatment step according to GINA guidelines
Treatment Patterns - Treatment adherence | From date of inclusion until the end of the study currently planned (2,5 years)
  Assessed using a Visual Analogue Scale (VAS) from 0 to 100, 0 means poor adherence and 100 good adherence
Treatment Patterns - Inhalation technique | From date of inclusion until the end of the study currently planned (2,5 years)
  Assessed by the clinician using national checklists
Subject's characteristics - Gender | From date of inclusion until the end of the study currently planned (2,5 years)
  Male/Female
Subject's characteristics - Marital status | From date of inclusion until the end of the study currently planned (2,5 years)
  Single, Married / De facto Union, Separated / Divorced, Widowed
Subject's characteristics - socio-economic and education level | From date of inclusion until the end of the study currently planned (2,5 years)
Subject's characteristics - occupational status | From date of inclusion until the end of the study currently planned (2,5 years)
Subject's characteristics - Smoking status & environmental tobacco smoke | From date of inclusion until the end of the study currently planned (2,5 years)
Subject's characteristics - Health related quality of life | From date of inclusion until the end of the study currently planned (2,5 years)
  Using EQ-5D. EQ-5D is a questionnaire which include five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). and is used to evaluate the quality of life. Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health).

CONTACTS AND LOCATIONS:
Overall Officials: João Fonseca, MD/PhD, Principal Investigator — cintesis; Jaime Correia de Sousa, MD/PhD, Principal Investigator — ICVS
Locations (31):
- Portugal (31):
  - Research Site, Alpendorada, Portugal
  - Research Site, Vila Cova Da Lixa, Portugal
  - Research Site, Aradas
  - Research Site, Arazede
  - Research Site, Braga
  - Research Site, Cascais
  - Research Site, Coimbra
  - Research Site, Evora
  - Research Site, Fafe
  - Research Site, Leiria
  - Research Site, Lisbon
  - Research Site, Mafra
  - Research Site, Montenegro
  - Research Site, Oeiras
  - Research Site, Ovar
  - Research Site, Pinhal Novo
  - Research Site, Ponte
  - Research Site, Porto
  - Research Site, Queluz
  - Research Site, Quinta Do Conde
  - Research Site, Ribeira de Pena
  - Research Site, Rio de Mouro
  - Research Site, Tavira
  - Research Site, Tomar
  - Research Site, Tondela
  - Research Site, Viana do Castelo
  - Research Site, Vila do Conde
  - Research Site, Vila Nova da Barquinha
  - Research Site, Vila Nova de Gaia
  - Research Site, Vila Real
  - Research Site, Vouzela

REFERENCES:
- [Derived] Jacome C, Brito D, Joao C, Lopes F, Santos J, Amorim L, Barbosa MJ, Pardal M, Teixeira P, Bernardo F, Fonseca JA, Correia-de-Sousa J. EPI-ASTHMA study protocol: a population-based multicentre stepwise study on the prevalence and characterisation of patients with asthma according to disease severity in Portugal. BMJ Open. 2022 Sep 19;12(9):e064538. doi: 10.1136/bmjopen-2022-064538. PMID 36123070
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2287R00155&attachmentIdentifier=97a5e988-7899-4336-9d93-4d32b4643f25&fileName=D2287R00155_(Epi-Asthma)_CSR_Synopsis_Portugal_03.03.2025.pdf&versionIdentifier=